CLINICAL TRIAL: NCT01940289
Title: Validation of Algometry for Use in the Human Foot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dundee Podiatry Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: PTM001
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Normative Algometric Pressures; Foot Pain
Keywords: algometry; pain; VAS
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- asymptomatic subjects attending podiatry clinic for nail care (Active Comparator): Algometric meter readings for perception of pain These subjects will have an algometric pressure threshold meter reading taken during their routine treatment visit to establish Algometric meter readings for perception of pain
  Interventions: Device: Algometric meter readings for perception of pain
- forefoot pain (Active Comparator): Algometric meter readings for perception of pain forefoot pain severity measured by both VAS and algometric pressure meter
  Interventions: Device: Algometric meter readings for perception of pain

INTERVENTIONS:
Device: Algometric meter readings for perception of pain
  Other Names: pressure threshold pain readings; pressure/pain readings

SUMMARY:
The primary aim is to examine whether there is a consistent range of pressure threshold values for the asymptomatic foot.Previous studies established the inter/intra-clinician reliability of pressure threshold measuring and have established a normative range of values within the trunk and upper body. Since the establishment of these values, pressure threshold testing has been used extensively in the head, neck, shoulders and spine as a clinical tool and a research aid. There has been little work using it in the lower limb and there are no guideline measurements for the clinician. By establishing a range of values for the foot,this study will enable the clinician to employ pressure threshold measuring as a clinical tool to easily and accurately identify areas of dysfunction and to objectively measure the effectiveness of treatment. It will allow the clinician to establish a degree of improvement or deterioration as it occurs in a patient's condition.

Secondary aims are to examine whether there is a correlation between visual analogue pain scale (VAS) scores and algometric pressure threshold scores for subjects with forefoot pain. This will help validate the tool for use in the foot. Since VAS is well documented and validated, this study will examine whether there is a correlation between VAS and algometry and whether there are gender or age differences in the range of measurements obtained. These areas have been addressed in previous studies but results have been contradictory and inconclusive and none of the previous studies focused on the foot.

An asymptomatic group of 384 subjects & symptomatic group of 160 subjects shall be selected from those attending a podiatric clinic for routine foot care who meet the inclusion criteria . Outcome me will be algometric pressure threshold testing, visual analogue pain scales and foot function index questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* All patients attending a local podiatric clinic for routine nail care or complaining of forefoot pain

Exclusion Criteria:

* forefoot surgery
* Diabetes
* Rheumatoid Arthritis
* Osteopenia
* All subjects with a diagnosed neurological condition
* Chronic pain at any body location
* Fibromyalgia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Algometric pressure threshold scores | 6 months
  Using algometric meter readings compared to Visual analogue pain scale readings to establish whether the two measures correlate

SECONDARY OUTCOMES:
visual analogue pain scale scores | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David G Cashley, BSc(Hons)Pod, Principal Investigator — Dundee Podiatry Clinic
Locations (1):
- Dundee Podiatry Clinic, Dundee, Angus, United Kingdom